CLINICAL TRIAL: NCT01626833
Title: Severe Decrease of Growth Velocity in Children With Anorexia Nervosa. Therapeutic Trial of Growth Hormone
Brief Title: Severe Decrease of Growth Velocity in Children With Anorexia Nervosa.Therapeutic Trial of Growth Hormone
Acronym: OREX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P090903; 2010-018560-16 (EudraCT Number)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Anorexia Nervosa; Interruption of Growth; Delayed Puberty; Osteopenia With Failure of Acquisition of Bone Mass
Keywords: anorexia nervosa; GH; Growth velocity
MeSH Terms: conditions — Anorexia Nervosa; Puberty, Delayed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOMATROPINE* : Norditropine® simplexx® (Active Comparator): SOMATROPINE* : Norditropine® simplexx®
  Interventions: Drug: SOMATROPINE* : Norditropine® simplexx®
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Drug: SOMATROPINE* : Norditropine® simplexx® — SOMATROPINE* : Norditropine® simplexx® - 15 mg/1,5 ml, injectable solution:Treatment with hGH is administered at a dose of 0.05 mg / kg / day (0.35 mg / kg / week) subcutaneously daily, preferably in the evening. The dose of hGH treatment will be adjusted according to weight gain, and reduced by 10% if the serum values of IGF-I SDS above 2.5 on 2 consecutive determinations at 3-month intervals are discovered by the biologist.
  Other Names: SOMATROPINE
  Arms: SOMATROPINE* : Norditropine® simplexx®
Biological: Placebo — Treatment with placebo is administered at a dose of 0.05 mg / kg / day (0.35 mg / kg / week) subcutaneously daily, preferably in the evening. The dose of placebo will be adjusted according to weight gain, and reduced by 10% if the serum values of IGF-I SDS above 2.5 on 2 consecutive determinations at 3-month intervals are discovered by the biologist.
  Arms: Placebo

SUMMARY:
Anorexia nervosa may be responsible for a catch- down or even an interruption of growth, delayed puberty and osteopenia with failure of acquisition of bone mass. The recovery of normal nutrition usually leads to a resumption of growth and pubertal development. However, despite a therapeutic nutritional and psychotherapeutic satisfactory approach, some patients have a significant short stature with reduced adult final height and a deficit of bone mass. The main objective is to evaluate the effect of growth hormone (hGH) treatment on the growth velocity in prepubertal children or children in early puberty with anorexia nervosa and significant reduction of height velocity. This is a single-center, controlled, randomized and double-blind clinical trial evaluating the efficacy of hGH treatment for 1 year against a placebo, on the growth velocity of prepubertal or children in early puberty with Anorexia nervosa and major catch-down.This period is followed by the evaluation of the hGH treatment in children receiving placebo and continued hGH treatment in the treatment arm for 1 year, in total 2 years of study for each child. This second period corresponds to an ethical consideration giving secondarily access to treatment for patients in the placebo group.

DETAILED DESCRIPTION:
Patients will be evaluated at baseline and at 3, 6, 9, 12, 15, 18, 21 and 24 months after the start of the trial. This evaluation will include a clinical evaluation and a biological (IGF-I, IGFBP-3, leptin, ghrelin, adiponectin, mineral metabolism, thyroid function, 24 hours urinary cortisol, as well as conventional electrolyte tolerance parameters), psychological and nutritional study body composition by absorptiometry at 0, 12 and 24 months. Evaluations will be conducted at the Center for Clinical Investigation at Hospital Robert Debre. The primary endpoint will be the linear growth rate 1 year after the start of the trial expressed in cm/1 year in the group with hGH compared to the placebo group. The secondary endpoints will be the height velocity expressed in SDS (standard deviation score), the data of body composition and psychological changes that will be assessed between the 2 arms at the end of the two years of the clinical trial. The data of body composition obtained by dual photon absorptiometry and biological data of mineral metabolism and growth factors are expressed in Z score compared to normal references that we have established in France, in healthy subjects according to age, gender and pubertal stage.

ELIGIBILITY:
Inclusion Criteria:

* Medical screening.
* Female and male subjects aged 8-16 years and 11 months, with clinical anorexia nervosa and / or reference to the diagnostic criteria of DSM-IV (1) before or at early puberty (Tanner stage 1 or 2) and with a prolonged Catch-Down for at least 18 months (HV ≤ 2 cm / year), with bone age ≤ 12 years in girls and ≤14 years in boys.
* Anorexia nervosa diagnosed at least 1 year before the study
* Growth velocity documented for at least 18 months before inclusion
* As with any child with a severe Catch-Down an assessment of GH secretion must be performed before inclusion (in the context of care) in the trial, which is not conditioned by the GH peak value : GH value of <20 miu / L will lead to the production of a brain MRI (in the context of care) that have to be normal (normal hypothalamic-pituitary axis and absence of tumor pathology) to allow Inclusion of the patient.
* Normal glucose tolerance
* Stable metabolic state with of weight gain of at least 10% of body weight from the time the body mass index was the lowest in relation to the occurrence of the disease and normal blood electrolytes (no hypokalemia) .
* Subjects whose holders have signed parental consent
* Subjects whose holders of parental authority are affiliated to a social security scheme
* CMU (CMU universal medical coverage).

Exclusion Criteria:

* Subjects in the mid-puberty (Tanner stage 3 or 4) or with menarche.
* Subjects with a chromosomal abnormality or other chronic disease associated chronic requiring long-term treatment.
* Impaired glucose tolerance or diabetes.
* Inability of the patient or the medical team to ensure the progress and monitoring under the protocol.
* Participation in another trial.
* Bradycardia ≤ 50 bpm.
* Children whose holders of parental authority are not beneficiaries of social security
* Contra-indication to SOMATROPINE

Ages: 8 Years to 203 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
the growth-velocity | 1 year
  the growth velocity will be evaluated 1 year after the start of the trial (cm/1an) compared between the group with the placebo and hGH

SECONDARY OUTCOMES:
growth-velocity | 2 years
  The secondary endpoints will be the growth-velocity expressed in SDS that will be assessed between the 2 arms at the end of the two years of clinical trial.
Body composition | 2 years
  The data of body composition that will be assessed between the 2 arms at the end of the two years of clinical trial. The data of body composition obtained by dual photon absorptiometry and biological data of mineral metabolism and growth factors are expressed in Z score compared to normal references that we have established in France, in healthy subjects according to age, gender and pubertal stage.
Psychological changes | 2 years
  Psychological changes that will be assessed between the 2 arms at the end of the two years of clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Leger Juliane, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France

REFERENCES:
- [Derived] Leger J, Fjellestad-Paulsen A, Bargiacchi A, Pages J, Chevenne D, Alison M, Alberti C, Guilmin-Crepon S. One Year of GH Treatment for Growth Failure in Children With Anorexia Nervosa: A Randomized Placebo-Controlled Trial. J Clin Endocrinol Metab. 2021 Jun 16;106(7):e2535-e2546. doi: 10.1210/clinem/dgab203. PMID 33772303